CLINICAL TRIAL: NCT02585414
Title: Assessment of Tear Film Thickness by Optical Coherence Tomography in Healthy Subjects and Subjects With Dry Eye Disease
Brief Title: Assessment of TFT by OCT in Healthy Subjects and Subjects With DES
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Other Study IDs: OPHT-070115
Record Dates: First submitted 2015-04-26; First posted 2015-10-23 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 85 healthy subjects with no history of DES
- 255 subjects with DES

SUMMARY:
Dry eye syndrome (DES) is a highly prevalent ocular condition with potential severe consequences for affected patients. DES can be either caused by decreased tear production or increased tear evaporation, both leading to an instable tear film. Despite many efforts, generally accepted methodologies to diagnose, assess the severity and monitor DES are still lacking. Moreover, widely used clinical methods such as tear break up time (BUT), fluorescein staining of the cornea or Schirmer test only poorly reflect patients´ complains.

One of the main problems in the diagnosis and treatment of DES is that the most critical component - the tear film itself - is difficult to characterize. The development of new ultra-high resolution optical coherence tomography systems allows now for the direct visualization of the human tear film and for the non-invasive in-vivo measurement of tear film thickness (TFT). The investigators could recently show that this system provides excellent reproducibility and is able to assess even subtle changes in TFT induced by therapeutic interventions. However, to which extent tear film thickness is associated with other standard clinical measures of DES is currently unknown. In the present study, the investigators set out to test the hypothesis that ocular TFT is a new and good surrogate parameter for the assessment of the severity of DES.

Consequently, the aim of the study presented in this protocol is to investigate whether and if so, to what extent clinical signs of DES and reported symptoms are reflected in ocular TFT. For this purpose, a cross sectional study in healthy subjects and patients with DES will be performed. This should allow the investigators to more specifically characterize the role of the tear film in DES and to assess whether measurement of TFT with OCT can be a promising surrogate parameter for the diagnosis and the follow up of DES.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy volunteers

* Men and women aged over 18 years
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 Dpt.

Inclusion criteria for patients with DES:

* Men and women aged over 18 years
* DES patients will be included based on three questions:

  * (1) "Have you ever been diagnosed (by a clinician) as having dry eye syndrome?"
  * (2) "Do you currently use artificial tear eyedrops or gel?"
  * (3) "For the past three months or longer, have you had dry eyes? (This is described as a foreign body sensation with itching and burning, sandy feeling, not related to allergy)."
* Normal ophthalmic findings except dry eye syndrome

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Wearing of contact lenses
* Intake of dietary supplements in the 3 months preceding the study
* History of glaucoma
* Treatment with corticosteroids in the 4 weeks preceding the study to topical treatment with any ophthalmic drug in the 4 weeks preceding the study (topical lubricants for patients with DES are allowed)
* Ocular infection or clinically significant inflammation
* Ocular surgery in the 3 months preceding the study
* Sjögren's syndrome
* Stevens-Johnson syndrome
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 85 healthy subjects with no history of DES 255 subjects with DES
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tear Film Thickness (TFT) as measured with Optical Coherence Tomography (OCT) | 1 month

SECONDARY OUTCOMES:
Tear Break Up Time | 1 month
Schirmer 1 test | 1 month
Corneal staining according to Oxford scale | 1 month
Tear osmolarity | 1 month
Ocular Surface Disease Index (OSDI) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Austria, Vienna, Austria